CLINICAL TRIAL: NCT02609425
Title: Intrathoracic Esophagogastric Anastomosis After Robot Assisted Minimally Invasive Esophagectomy Using STRATAFIX
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, loay kabbani, MD, Vice Chair of Clinical Research, Surgery, Henry Ford Health System
Other Study IDs: Esophagogastric Anastomosis
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- STRATAFIX: Anastomosis of esophagus to stomach
  Interventions: Device: Stratafix PGA Suture

INTERVENTIONS:
Device: Stratafix PGA Suture — Subject leak Stricture rates post procedure

SUMMARY:
Determine the safety and efficacy of novel suture in esophageal anastomosis. Specific Aims: 1) Determine the safety of using STRATAFIX suture in esophagogastric anastomosis by measuring anastomotic leak rate; and 2) Determine efficacy of STRATAFIX suture in esophagogastric anastomosis by measure anastomotic stricture rate.

DETAILED DESCRIPTION:
The purpose of the proposed study is to demonstrate that a hand sewn anastomosis using STRATAFIX is safe and effective after minimally invasive esophagectomy and capture anastomotic leak and stricture rate after esophagectomy. If proven, one may reasonably conclude that STRATAFIX may be safely used in other less complex anastomoses and closures throughout the gastrointestinal tract. Furthermore, the work may promote the utilization of STRATAFIX for other applications, e.g. closure of the vaginal cuff after hysterectomy. The study is proposed to demonstrate the safety and efficacy of utilizing an absorbable running suture for completion of a hand swen intra thoracic esophago-gastric anastomosis during minimally invasive esophagectomy. There are many advantages to hand sewn anastomosis compared with stapled, e.g. EEA anastomosis. Two potential advantages are a lower leak rate and a lower stricture rate. Currently hand swen anastomosis is performed with interrupted suture of absorbable material. While effective, this technique requires multiple sutures, thus increasing operative time and material cost. Utilizing a running suture technique has the potential to reduce operative time and overall operative cost. Furthermore, it may lead to a reduction in postoperative morbidity by reducing anastomotic leak rate and structure formation. The hypothesis of the protocol is to evaluate the use of STRATAFIX in performing a hand swen intrathoracic anastomosis after minimally invasive esophagectomy is non inferior (and may be superior) to historical cases in which the anastomosis was completed using other types of suture material. Inclusion criteria: (1) All patients with esophageal cancer who are deemed candidates for minimally invasive robot assisted Ivor Lewis esophagogastrectomy. (2) Patients who provide written informed consent for the study. Exclusion criteria: Standard minimally invasive esophagectomy technique will be employed. (1) Creation of gastric conduit laparoscopically. (2) Robotic assisted esophageal mobilization through the right chest. (3) Robotic assisted intrathoracic anastomosis at or above the level of the azygous vein. (4) Barium swallow performed on post operative day 5-7 to assess anastomotic integrity. (5) Periodic clinical follow up on an outpatient basis to assess need for any interventions for anastomotic stricture.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with esophageal cancer who are deemed candidates for minimally invasive robot assisted Ivor Lewis esophagogastrostomy.
2. Patients who provide written informed consent for the study.

Exclusion Criteria:

1. Any patient with esophageal cancer who is not deemed a surgical candidate or who is not deemed a candidate for the Ivor Lewis technique of esophagectomy (with intrathoracic anastomosis).
2. Any patient less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with esophageal cancer undergoing a planned minimally invasive robot assisted Ivor Lewis esophagogastrostomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zane Hammoud, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Cerfolio RJ, Bryant AS, Hawn MT. Technical aspects and early results of robotic esophagectomy with chest anastomosis. J Thorac Cardiovasc Surg. 2013 Jan;145(1):90-6. doi: 10.1016/j.jtcvs.2012.04.022. Epub 2012 Aug 19. PMID 22910197
- [Background] Sarkaria IS, Rizk NP, Finley DJ, Bains MS, Adusumilli PS, Huang J, Rusch VW. Combined thoracoscopic and laparoscopic robotic-assisted minimally invasive esophagectomy using a four-arm platform: experience, technique and cautions during early procedure development. Eur J Cardiothorac Surg. 2013 May;43(5):e107-15. doi: 10.1093/ejcts/ezt013. Epub 2013 Jan 30. PMID 23371971

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participipants: All patients enrolled on the study.
Period: Overall Study
Arm/Group | All Participipants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All patients enrolled on the study
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 25
  African American | 2
  Hispanic | 3
Region of Enrollment: United States [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Anastomotic Leak Rate After Esophagectomy
Description: Analysis specific to anastomosis leak will be analyzed and compared with historically published results to determine whether Stratafix suture is appropriate in this application.
Time Frame: 5-7 Days to assess anastomotic integrity
Population: Data were not collected
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Anastomotic Stricture Rate After Esophagectomy
Description: Analysis specific to anastomosis stricture will be analyzed and compared with historically published results to determine whether Stratafix suture is appropriate in this application.
Time Frame: 5-7 days to assess anastomotic integrity
Population: Data were not collected
Arm/Group | All Participipants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months after surgery date
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT02609425/Prot_000.pdf